CLINICAL TRIAL: NCT02294825
Title: The North-West Inter Regional Female Cohort for Patients With Endometriosi
Brief Title: The North-West Inter Regional Female Cohort for Patients With Endometriosis
Acronym: CIRENDO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Rouen (Other)
Collaborators: University Hospital, Lille (Other); University Hospital, Caen (Other); Amiens University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2009-099-HP
Record Dates: First submitted 2014-11-16; First posted 2014-11-19 (Estimated); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Endometriosis
Keywords: deep endometriosis;; colorectal endometriosis; surgery; medical treatment; fertility
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: various surgical procedures in endometriosis — Shaving, disc excision and colorectal resection; ureterolysis or ureter resection; bladder resection; ablation of endometriomas using plasma energy; excision and ablation of deep and superficial lesions

SUMMARY:
All women managed for endometriosis are included and followed up through the CIRENDO database.

Information is obtained from surgical and histological records and from self-questionnaires completed before surgery. Standardized gastrointestinal questionnaires (KESS, GIQLI, WEXNER, FIQL and Bristol) are routinely used to assess bowel function. Data recording, patient contact and follow-up are carried out by a clinical research technician. Postoperative follow-up is based on data from the afore-mentioned questionnaires completed at 1, 3, 5 and 7 years.

DETAILED DESCRIPTION:
All women managed for endometriosis are included and followed up through the CIRENDO database (the North-West Inter Regional Female Cohort for Patients with Endometriosis), a prospective cohort financed by the G4 Group (The University Hospitals of Rouen, Lille, Amiens and Caen), and coordinated by the principal investigator (H.R.). Information is obtained from surgical and histological records and from self-questionnaires completed before surgery. Standardized gastrointestinal questionnaires (KESS, GIQLI, WEXNER, FIQL and Bristol) are routinely used to assess bowel function. Data recording, patient contact and follow-up are carried out by a clinical research technician. Women are included in the CIRENDO database only when endometriosis is confirmed by both surgical exploration and biopsy. Postoperative follow-up is based on data from the afore-mentioned questionnaires completed at 1, 3, 5 and 7 years. Prospective data recording and analysis were approved by the French authorities CNIL (Commission Nationale de l'Informatique et des Libertés) and CCTIRS (Comité Consultatif pour le Traitement de l'Information en matière de Recherche dans le domaine de la Santé).

ELIGIBILITY:
Inclusion Criteria:

* Endometriosis revealed on histological specimens

Exclusion Criteria:

* None

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients surgically managed for endometriosis in one of centers involved in the study
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2009-06; Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Recurrences | 7 years
  rate of recurrences at 1,3,5 and 7 years postoperatively

SECONDARY OUTCOMES:
Risk factors for endometriosis | 1 year
  Association of various antecedents with specific localizations of features of the endometriosis
Digestive functional outcomes | 7 years
  Bowel function in patients managed for bowel endometriosis by various procedures
Fertility | 7 years
  Rate of pregnancy at 1, 3, 5, and 7 years postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Horace Roman, Principal Investigator — University Hospital, Rouen
Locations (1):
- Clinique Gynécologique et Obstétricale, Rouen, France

REFERENCES:
- [Result] Roman H, Bubenheim M, Auber M, Marpeau L, Puscasiu L. Antimullerian hormone level and endometrioma ablation using plasma energy. JSLS. 2014 Jul-Sep;18(3):e2014.00002. doi: 10.4293/JSLS.2014.00002. PMID 25392649
- [Result] Roman H, Auber M, Bourdel N, Martin C, Marpeau L, Puscasiu L. Postoperative recurrence and fertility after endometrioma ablation using plasma energy: retrospective assessment of a 3-year experience. J Minim Invasive Gynecol. 2013 Sep-Oct;20(5):573-82. doi: 10.1016/j.jmig.2013.02.016. Epub 2013 Jun 10. PMID 23759693
- [Result] Roman H, Ness J, Suciu N, Bridoux V, Gourcerol G, Leroi AM, Tuech JJ, Ducrotte P, Savoye-Collet C, Savoye G. Are digestive symptoms in women presenting with pelvic endometriosis specific to lesion localizations? A preliminary prospective study. Hum Reprod. 2012 Dec;27(12):3440-9. doi: 10.1093/humrep/des322. Epub 2012 Sep 7. PMID 22962316
- [Result] Rozsnyai F, Roman H, Resch B, Dugardin F, Berrocal J, Descargues G, Schmied R, Boukerrou M, Marpeau L; CIRENDO Study Group. Outcomes of surgical management of deep infiltrating endometriosis of the ureter and urinary bladder. JSLS. 2011 Oct-Dec;15(4):439-47. doi: 10.4293/108680811X13176785203798. PMID 22643496
- [Result] Bridoux V, Roman H, Kianifard B, Vassilieff M, Marpeau L, Michot F, Tuech JJ. Combined transanal and laparoscopic approach for the treatment of deep endometriosis infiltrating the rectum. Hum Reprod. 2012 Feb;27(2):418-26. doi: 10.1093/humrep/der422. Epub 2011 Dec 8. PMID 22158086
- [Result] Auber M, Bourdel N, Mokdad C, Martin C, Diguet A, Marpeau L, Roman H. Ultrasound ovarian assessments after endometrioma ablation using plasma energy. Fertil Steril. 2011 Jun 30;95(8):2621-4.e1. doi: 10.1016/j.fertnstert.2011.04.090. Epub 2011 May 31. PMID 21621773
- [Result] Vassilieff M, Suaud O, Collet-Savoye C, Da Costa C, Marouteau-Pasquier N, Belhiba H, Tuech JJ, Marpeau L, Roman H. [Computed tomography-based virtual colonoscopy: an examination useful for the choice of the surgical management of colorectal endometriosis]. Gynecol Obstet Fertil. 2011 Jun;39(6):339-45. doi: 10.1016/j.gyobfe.2011.04.004. Epub 2011 May 18. French. PMID 21596608
- [Result] Roman H, Pura I, Tarta O, Mokdad C, Auber M, Bourdel N, Marpeau L, Sabourin JC. Vaporization of ovarian endometrioma using plasma energy: histologic findings of a pilot study. Fertil Steril. 2011 Apr;95(5):1853-6.e1-4. doi: 10.1016/j.fertnstert.2010.11.038. Epub 2010 Dec 17. PMID 21168130
- [Derived] Badescu A, Roman H, Barsan I, Soldea V, Nastasia S, Aziz M, Puscasiu L, Stolnicu S. Patterns of Bowel Invisible Microscopic Endometriosis Reveal the Goal of Surgery: Removal of Visual Lesions Only. J Minim Invasive Gynecol. 2018 Mar-Apr;25(3):522-527.e9. doi: 10.1016/j.jmig.2017.10.026. Epub 2017 Oct 31. PMID 29097234
- [Derived] Darwish B, Stochino-Loi E, Pasquier G, Dugardin F, Defortescu G, Abo C, Roman H. Surgical Outcomes of Urinary Tract Deep Infiltrating Endometriosis. J Minim Invasive Gynecol. 2017 Sep-Oct;24(6):998-1006. doi: 10.1016/j.jmig.2017.06.005. Epub 2017 Jun 15. PMID 28624664
- [Derived] Roman H, Darwish B, Bridoux V, Chati R, Kermiche S, Coget J, Huet E, Tuech JJ. Functional outcomes after disc excision in deep endometriosis of the rectum using transanal staplers: a series of 111 consecutive patients. Fertil Steril. 2017 Apr;107(4):977-986.e2. doi: 10.1016/j.fertnstert.2016.12.030. Epub 2017 Jan 27. PMID 28139235
- [Derived] Roman H, Hennetier C, Darwish B, Badescu A, Csanyi M, Aziz M, Tuech JJ, Abo C. Bowel occult microscopic endometriosis in resection margins in deep colorectal endometriosis specimens has no impact on short-term postoperative outcomes. Fertil Steril. 2016 Feb;105(2):423-9.e7. doi: 10.1016/j.fertnstert.2015.09.030. Epub 2015 Oct 29. PMID 26474734